CLINICAL TRIAL: NCT03324841
Title: Caris Molecular Intelligence® and Caris Centers of Excellence for Precision Medicine NetworkTM Outcomes Associated Repository
Brief Title: POA Prospective Repository
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Caris Science, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: COE-001-0815
Record Dates: First submitted 2017-10-13; First posted 2017-10-30 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Solid Tumor, Adult; Oncology
Keywords: Molecular Profiling; Biomarker Analysis; Next Generation Sequencing
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MI Profiling: Subjects must have undergone Caris MI Profiling in order to be eligible for the study. No required intervention is dictated by the protocol.
  Interventions: Diagnostic Test: Caris MI Profiling

INTERVENTIONS:
Diagnostic Test: Caris MI Profiling — Customized comprehensive biomarker testing

SUMMARY:
This repository is a multi-center, outcomes study designed to collect data on the demographics, presentation, diagnosis, treatment, cost of associated care, quality of life, and outcomes of subjects utilizing Caris Molecular Intelligence® (CMI) Services for the treatment of cancer.

DETAILED DESCRIPTION:
This repository is a multi-center, outcomes study designed to collect data on the demographics, presentation, diagnosis, treatment, cost of associated care, quality of life, and outcomes of subjects utilizing Caris Molecular Intelligence® (CMI) Services for the treatment of cancer. Prior to enrolling a subject, the subject's physician will have made the independent decision whether or not to utilize the drug associations provided by CMI and made clinical treatment choices as appropriate. Thus, data captured and reported provides a "real world" perspective on diagnosis, treatment, cost, and outcomes.

Prospective data will be obtained only from consented patients or patients who have died or have been lost to follow-up. Lost to follow-up is defined as a subject who has not returned for continued care or evaluation (e.g., disability, relocation or unresponsiveness). Site coordinators are required attempt to contact the subject 3 times before deeming them lost to follow up. Data collection and the protection of privacy are discussed in the Methods section below.

In addition to treatment and response data, initial diagnosis and staging results will be recorded as well as any recurrence information. As the investigators are capturing the subject's cancer treatment as a whole, results from pertinent cancer-related tests performed by outside entities for eligible subjects will need to be collected by the site coordinator and maintained at the site accordingly for reporting and monitoring purposes.

ELIGIBILITY:
Inclusion Criteria:

* Subject's age must be greater than or equal to 18 years and must have received CMI testing

Exclusion Criteria:

* Due to the complexity of state and federal requirements governing the participation of prisoners in research, prisoners-patients shall not be approached for participation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects who received Caris MI Profiling at one of the Precision Oncology Alliance (POA) sites
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-06-07 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Effecting Change | within 5 years
  Effecting change in disease treatment processes by advancing precision medicine and improving care for cancer through acquiring and sharing valuable molecular tumor profiling information and clinical outcomes in a collaborative, secure environment.
Performing retrospective research | within 5 years
  Performing retrospective research including clinical presentation, treatment and outcomes. This eligible cohort includes select subjects who have already undergone Caris Molecular Intelligence® evaluation for diagnosis and/or treatment management.
Evaluate the frequency of specific clinical events | within 5 years
  Evaluate the frequency of specific clinical events in relation to risk factors, diagnosis and treatments provided via the collection of outcomes data through automated data capture systems provided by a third-party data entity and manually-entered data when needed.
Provide information access that is vital to research collaborators | within 5 years
  Provide information access that is vital to research collaborators, including potential researchers from pharmaceutical companies, governmental agencies, academia, healthcare providers, and payors, with catalogued subject outcome data for the use of drug development discoveries, clinically relevant research trials, publications and posters, the implementation of future healthcare policies, characterization of trends in practice patterns and their relation to subject outcomes and the economic impact of differing evaluation, treatment, and management paradigms.
Cultivate a repository for assay development | within 5 years
  Cultivate a repository for assay development and validation of emerging technologies to enhance clinical cancer care.

CONTACTS AND LOCATIONS:
Overall Officials: W. Michael Korn, MD, Study Director — Caris Life Sciences
Locations (11):
- United States (11):
  - HonorHealth, Scottsdale, Arizona
  - University of Arizona, Tucson, Arizona
  - St. Joseph Heritage Healthcare, Irvine, California
  - John Wayne Cancer Institute, Santa Monica, California
  - MedStar Health Research Institute, Inc., Washington D.C., District of Columbia
  - AdventHealth Orlando Cancer Institute, Orlando, Florida
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - University of Cincinnati Health, LLC, Cincinnati, Ohio
  - The Institute for Cancer Research dba The Research Institute of Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - The West Clinic, Germantown, Tennessee
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas